CLINICAL TRIAL: NCT01270425
Title: Sonographic Characterization of the Thyroid Gland in Patients With Systemic Sclerosis With and Without Hashimoto Thyroiditis
Brief Title: Sonographic and Laboratory Evaluation of the Thyroid Gland in Patients With Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC11175-10CTIL
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2012-03

CONDITIONS: Systemic Sclerosis; Hashimoto Thyroiditis; Thyroid Nodules
Keywords: systemic sclerosis; hashimoto thyroiditis; thyroid nodules
MeSH Terms: conditions — Scleroderma, Systemic; Hashimoto Disease; Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Systemic sclerosis (SSc) is a systemic disease that involves various organs such as the skin, kidneys, gastrointestinal tract and lungs. Dysfunction of the thyroid gland is prevalent in these patients and may be related to thyroid fibrosis or to thyroid autoimmune disease, i.e. hashimoto's thyroiditis. Thyroid nodules are prevalent in the general population, although some reports suggest they might be more frequent in patients with SSc. Hashimoto's thyroiditis, by itself, carries a higher risk for thyroid nodules and thyroid cancer.

The aim of the study:To characterize sonographycally the thyroid gland of patients with SSc with and without Hashimoto's disease

DETAILED DESCRIPTION:
The study protocol Fifty patients with SSc according to the current international classification will be included in the study. The patients, followed-up regularly in an out-patient clinic, will be tested for their thyroid function tests as well as the presence of thyroid auto antibodies. Clinical data will be collected from their medical records. Ultrasonographic examination of the thyroid gland will be performed by a single examiner. The gland will be characterized in detail with regards to its size and echotexture and cervical lymph nodes will be detected. The number and size of its nodules will be described as well as their echoic pattern (iso, hyperechoic or hypoechoic) calcifications (micro and macro), and borders status. Large nodules (≥ 1 cm in diameter) or with malignancy- associated characteristics will be aspirated according to current clinical practice. Treatment will be given according to the cytology diagnosis. Thyroid hormone supplementation will be recommended when thyrotropin level >8 mIU/L or according to clinical judgment of the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of systemic sclerosis

Exclusion Criteria:

* non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SSc according to the current international classification
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
There are no spesific outcome measures from trail | Nnone
  the measures from trail are equal to vast population

CONTACTS AND LOCATIONS:
Overall Officials: Pnina Rotman-Pikielny, MD, Principal Investigator — Meir Medical Center, Israel
Locations (1):
- Meir Medical Center, Kfar Saba, Israel